CLINICAL TRIAL: NCT01164215
Title: Multicenter Study Investigating Utilization of Pharmacokinetic-Guided 5-Fluorouracil in Patients Receiving mFOLFOX6 With or Without Bevacizumab
Brief Title: Biomarker-Guided Fluorouracil in Treating Patients With Colorectal Cancer Receiving Combination Chemotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 0918; P30CA016086 (NIH); CDR0000681338 (Other: PDQ number)
Record Dates: First submitted 2010-07-15; First posted 2010-07-16 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: Colorectal Cancer; Diarrhea; Neutropenia
Keywords: neutropenia; diarrhea; stage I colon cancer; stage II colon cancer; stage III colon cancer; stage IV colon cancer; recurrent colon cancer; stage I rectal cancer; stage II rectal cancer; stage III rectal cancer; stage IV rectal cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Diarrhea; Neutropenia; Colonic Neoplasms; Rectal Neoplasms | interventions — Fluorouracil; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- mFOLFOX6 (Experimental): Patients will receive cycle 1 of standard dose mFOLFOX6, with the same dose of mFOLFOX6 continued in subsequent cycles, once patient achieves the target AUC.
  mFOLFOX 6 is a regimen comprised of Oxaliplatin + Leucovorin +5-Fluorouracil (FU)
  Interventions: Drug: fluorouracil; Drug: leucovorin; Drug: oxaliplatin

INTERVENTIONS:
Drug: fluorouracil — 200-400 mg/m2 intravenously, 1 -5 minutes, once every 2 weeks 2400 mg/m2 intravenously over a period of 46 hours, once every 2 weeks
  Other Names: 5FU
Drug: leucovorin — 200-400 mg/m2, intravenously over a period of 2 hours, once every 2 weeks
  Other Names: leucovorin calcium
Drug: oxaliplatin — 85 mg/m2, intravenously for 2 hours, once every 2 weeks
  Other Names: Eloxatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fluorouracil, oxaliplatin, and leucovorin calcium, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug, combination chemotherapy, may kill more tumor cells. Studying samples of blood in the laboratory from patients with cancer receiving fluorouracil in combination with oxaliplatin and leucovorin calcium may help doctors learn how fluorouracil works in the body and how patients will respond to treatment.

PURPOSE: This phase I trial is studying biomarker-guided fluorouracil in treating patients with colorectal cancer receiving combination chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine whether 4 courses of pharmacokinetic (PK)-guided 5-fluorouracil chemotherapy improves the ability to achieve a targeted area under the curve (20 to 25 mg*hr/L) in patients with colorectal cancer receiving mFOLFOX6 chemotherapy as compared to historical non-PK-guided therapy in patients treated with a similar FOLFOX regimen.

Secondary

* To determine and compare the incidence of neutropenia and diarrhea in patients treated with these regimens.

OUTLINE: This is a multicenter study.

* Standard mFOLFOX6 (course 1): Patients receive fluorouracil IV bolus over 1-5 minutes followed by fluorouracil IV continuously over 46 hours, oxaliplatin IV over 2 hours, and leucovorin calcium IV over 2 hours on day 1.

Patients undergo plasma sample collection periodically during study for pharmacokinetic (PK)-guided fluorouracil dose determination for courses 2-4.

* PK-guided mFOLFOX6 (courses 2-4): Patients receive fluorouracil bolus, oxaliplatin, and leucovorin calcium as in course 1. Patients also receive fluorouracil* IV continuously as determined by the PK-guided analysis.

NOTE: *The continuous infusion fluorouracil dose adjustment is calculated based on the results of PK plasma concentrations and the corresponding AUC from the preceding course.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed colorectal cancer
* Patients scheduled to receive mFOLFOX6 (in the adjuvant setting or for metastatic disease) as part of their chemotherapy regimen

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 6 months
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Serum creatinine ≤ 1.5 mg/dL
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN (≤ 5 times ULN in the presence of liver metastases)
* Fertile patients must use effective contraception
* Negative pregnancy test
* Not pregnant or nursing
* No serious concomitant systemic disorders, including active infection that, in the opinion of the investigator, would compromise the patient's safety or ability to complete the study
* No altered mental status precluding understanding of the informed consent process and/or completion of the necessary studies
* Must be able to follow protocol requirements and give informed consent

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Concurrent bevacizumab allowed
* No concurrent warfarin (Coumadin®)

  * Concurrent enoxaparin (Lovenox®) allowed
* No concurrent theophylline or aminophylline
* No chocolate beginning 12 hours before day 1 of each course and through the end of that course's fluorouracil continuous IV

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2010-02; Primary Completion 2012-11 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Achievement of targeted AUC using pharmacokinetic (PK)-guided 5 fluorouracil as part of mFOLFOX6 therapy | During first 4 cycles of drug therapy

SECONDARY OUTCOMES:
Toxicity differences between PK-guided therapy versus non-PK-guided therapy | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Christine M. Walko, PharmD, BCOP, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (5):
- United States (5):
  - Cancer Care of Western North Carolina, Asheville, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - Leo W. Jenkins Cancer Center at ECU Medical School, Greenville, North Carolina
  - Rex Cancer Center at Rex Hospital, Raleigh, North Carolina
  - Marion L. Shepard Cancer Center, Washington, North Carolina

REFERENCES:
- [Derived] Williams GR, Deal AM, Shachar SS, Walko CM, Patel JN, O'Neil B, McLeod HL, Weinberg MS, Choi SK, Muss HB, Sanoff HK. The impact of skeletal muscle on the pharmacokinetics and toxicity of 5-fluorouracil in colorectal cancer. Cancer Chemother Pharmacol. 2018 Feb;81(2):413-417. doi: 10.1007/s00280-017-3487-2. Epub 2017 Nov 20. PMID 29159476
- [Derived] Patel JN, O'Neil BH, Deal AM, Ibrahim JG, Sherrill GB, Olajide OA, Atluri PM, Inzerillo JJ, Chay CH, McLeod HL, Walko CM. A community-based multicenter trial of pharmacokinetically guided 5-fluorouracil dosing for personalized colorectal cancer therapy. Oncologist. 2014 Sep;19(9):959-65. doi: 10.1634/theoncologist.2014-0132. Epub 2014 Aug 12. PMID 25117066